CLINICAL TRIAL: NCT01327053
Title: Phase II, Randomized Double-blind Study of Efficacy and Safety of Two Dose Levels of LDE225 in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Brief Title: A Phase II Study of Efficacy and Safety in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Acronym: BOLT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDE225A2201; 2010-022629-14 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Basal Cell Carcinoma
Keywords: locally advanced basal cell carcinoma; metastatic basal cell carcinoma; LDE225; sonidegib; Basel Cell Carcinoma (BCC); skin cancer; Basel Cell Carcinoma; BCC
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — sonidegib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LDE225 200 mg (Experimental): The study was double blinded and enrolled at least 50 evaluable patients in the 200 mg LDE225 arm. The efficacy and safety of LDE225 was analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 200 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
  Interventions: Drug: LDE225
- LDE225 800 mg (Experimental): The study was double blinded and enrolled at least 100 evaluable patients in the 800 mg LDE225 arm. The efficacy and safety of LDE225 was analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 800 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225 was administered orally, on a continuous once daily dosing schedule and was supplied as 200 mg hard gelatin capsules in bottles. Every 4 weeks on the day of study visit, patients received a prescription of an adequate drug supply for self-administration at home. The 800 mg dose patients received 4 capsules of LDE225 and 200 mg dose arm patients received 1 LDE225 capsule + 3 placebo capsules.
  Other Names: Sonidegib

SUMMARY:
This study assessed the efficacy and safety of oral treatment with two dose levels of LDE225 in patients with locally advanced or metastatic BCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced BCC and metastatic BCC
* Patients with adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Patients who had had major surgery within 4 weeks of initiation of study medication
* Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract, or known malabsorption syndromes.
* Patients with concurrent medical conditions that may interfere or potentially affect the interpretation of the study.
* Patients with neuromuscular disorders or are on concurrent treatment with drugs that may cause muscle damage.
* Patients who were on concurrent therapy with other anti-neoplastic agents.
* Patients who had taken part in an experimental drug within 4 weeks of initiation of study medication.
* Pregnant or nursing (lactating) women
* Women of child bearing potential unwilling to use 2 forms of highly effective contraception throughout the study and for 3 months after the last treatment
* Fertile males not willing to use condoms throughout the study and for 3 months after the last treatment.
* Patients who were unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2013-06-28 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (22):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California at Los Angeles UCLA 3, Los Angeles, California
  - Stanford University Medical Center Stanford Univ 2, Stanford, California
  - University of Colorado School of Medicine UC, Aurora, Colorado
  - Washington Hospital Center Wash Hospital, Washington D.C., District of Columbia
  - H Lee Moffitt Cancer Center and Research Institute Cutaneous Onc Dept, Tampa, Florida
  - NorthwesternUniv.Med.School/Robert H. Lurie Comp.Cancer Ctr Study coordinator, Chicago, Illinois
  - Dana Farber Cancer Institute DFCI - MA, Boston, Massachusetts
  - Henry Ford Hospital Henry Ford, Detroit, Michigan
  - Washington University School Of Medicine-Siteman Cancer Ctr Siteman, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada CCC of Nevada- Southwest (2), Las Vegas, Nevada
  - Hackensack University Medical Center Hackensack (SC), Hackensack, New Jersey
  - New York University Medical Center SC-2, New York, New York
  - Penn State University / Milton S. Hershey Medical Center Hershey Medical, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center UPMC, Pittsburgh, Pennsylvania
  - Baylor Health Care System/Sammons Cancer Center Baylor Texas Oncology, Dallas, Texas
  - Texas Oncology Tex Onc 3, Dallas, Texas
  - Texas Oncology Texas Onc - Amarillo, Dallas, Texas
  - University of Texas MD Anderson Cancer Center MD Anderson, Houston, Texas
  - Texas Oncology Cancer Care & Research Center, Waco, Texas
  - Texoma Cancer Center Texoma Cancer Center, Wichita Falls, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman/Univ UT, Salt Lake City, Utah
- Australia (2):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Geelong, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Wilrijk
- Canada (2):
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
- France (5):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stade
- Novartis Investigative Site, Athens, Greece
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Italy (2):
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich
- United Kingdom (7):
  - Novartis Investigative Site, High Heaton, Newcastle Upon Tyne
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gutzmer R, Robert C, Loquai C, Schadendorf D, Squittieri N, Arntz R, Martelli S, Dummer R. Assessment of various efficacy outcomes using ERIVANCE-like criteria in patients with locally advanced basal cell carcinoma receiving sonidegib: results from a preplanned sensitivity analysis. BMC Cancer. 2021 Nov 19;21(1):1244. doi: 10.1186/s12885-021-08968-1. PMID 34798846
- [Derived] Lewis K, Dummer R, Farberg AS, Guminski A, Squittieri N, Migden M. Effects of Sonidegib Following Dose Reduction and Treatment Interruption in Patients with Advanced Basal Cell Carcinoma During 42-Month BOLT Trial. Dermatol Ther (Heidelb). 2021 Dec;11(6):2225-2234. doi: 10.1007/s13555-021-00619-4. Epub 2021 Oct 20. PMID 34669179
- [Derived] Lear JT, Migden MR, Lewis KD, Chang ALS, Guminski A, Gutzmer R, Dirix L, Combemale P, Stratigos A, Plummer R, Castro H, Yi T, Mone M, Zhou J, Trefzer U, Kaatz M, Loquai C, Kudchadkar R, Sellami D, Dummer R. Long-term efficacy and safety of sonidegib in patients with locally advanced and metastatic basal cell carcinoma: 30-month analysis of the randomized phase 2 BOLT study. J Eur Acad Dermatol Venereol. 2018 Mar;32(3):372-381. doi: 10.1111/jdv.14542. Epub 2017 Nov 6. PMID 28846163
- [Derived] Migden MR, Guminski A, Gutzmer R, Dirix L, Lewis KD, Combemale P, Herd RM, Kudchadkar R, Trefzer U, Gogov S, Pallaud C, Yi T, Mone M, Kaatz M, Loquai C, Stratigos AJ, Schulze HJ, Plummer R, Chang AL, Cornelis F, Lear JT, Sellami D, Dummer R. Treatment with two different doses of sonidegib in patients with locally advanced or metastatic basal cell carcinoma (BOLT): a multicentre, randomised, double-blind phase 2 trial. Lancet Oncol. 2015 Jun;16(6):716-28. doi: 10.1016/S1470-2045(15)70100-2. Epub 2015 May 14. PMID 25981810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization was stratified across the two treatment arms according to the stage of disease (laBCC or mBCC), histological subtype (non-aggressive or aggressive for laBCC patients) and the regions (Australia, Europe, and North America).
Pre-assignment Details: All eligible, enrolled patients were randomized in 1:2 ratio to sonidegib treatment with either 200 mg or 800 mg once-daily dose. In total, 230 patients were evaluated as FAS population: 79 and 151 patients randomized to 200mg and 800 mg sonidegib respectively. However, 1 patient randomized to 800 mg sonidegib did not receive study treatment.
Groups:
- LDE225 (Sonidegib) 200 mg: The study is double blinded and will enroll at least 50 evaluable patients in the 200 mg LDE225 arm. The efficacy and safety of LDE225 will be analyzed separately in each group. Patients who meet all the inclusion and none of the exclusion criteria will be treated with 200 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
- LDE225 (Sonidegib) 800 mg: The study is double blinded and will enroll at least 100 evaluable patients in the 800 mg LDE225 arm. The efficacy and safety of LDE225 will be analyzed separately in each group. Patients who meet all the inclusion and none of the exclusion criteria will be treated with 800 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
Period: Overall Study
Arm/Group | LDE225 (Sonidegib) 200 mg | LDE225 (Sonidegib) 800 mg
Started | 79 | 151
Untreated | 0 | 1 (one patient randomized to LDE225 (sonidegib) 800 mg did not receive study treatment)
Patients Cont. to Next Phase of Trial | 52 | 89
Survival Follow-up | 33 | 49
Post-treatment Follow-up | 19 | 40
Completed | 0 | 0
Not Completed | 79 | 151
Not completed — Adverse Event | 23 | 57
Not completed — Patient/guardian decision | 11 | 35
Not completed — Physician Decision | 10 | 14
Not completed — Death | 1 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Non-compliance with study treatment | 0 | 5
Not completed — Study terminated by Sponsor | 1 | 3
Not completed — Progressive disease | 31 | 26
Not completed — Protocol Violation | 0 | 1
Not completed — Untreated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all patients who were assigned study treatment irrespective of receiving it (all randomized patients). Patients were classified according to the treatment they were assigned in accordance with the intention-to-treat (ITT) principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225 (Sonidegib) 200 mg | LDE225 (Sonidegib) 800 mg | Total
Number analyzed (Participants) | 79 | 151 | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (15.67) | 63.6 (14.59) | 64.3 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 55 | 86
  Male | 48 | 96 | 144
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 0 | 1 | 1
  Caucasian | 71 | 145 | 216
  Other | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Central Review According to mRECIST (for Locally Advanced Basal Cell Carcinoma (laBCC)) and RECIST 1.1 (for Metastatic Basal Cell Carcinoma (mBCC)) Per Primary Efficacy Analysis Set (pEAS)
Description: ORR is the percentage of patient's objective response (ORR) by 6 months after starting LDE225 treatment. A responder was defined as a subject with confirmed partial response (PR) or confirmed complete response (CR) 6 months after starting LDE225 treatment.Treatment with sonidegib was considered sufficiently efficacious if the observed ORR on any treatment arm at the end of the study was 30% or higher. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 6 months
Population: The primary efficacy analysis set (pEAS) was a subset of the full analysis set (FAS) including patients with laBCC with tumors that were adequately assessed by MRI or photography or both, & including all patients with mBCC included in the FAS which comprised all patients who were assigned study treatment irrespective of receiving it.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- LDE225 200mg laBCC: The efficacy and safety of LDE225 200mg laBCC cohort were analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 200 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
- LDE225 800mg laBCC: The efficacy and safety of LDE225 800mg laBCC cohort were analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 800 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
- LDE225 200mg mBCC: The efficacy and safety of LDE225 200mg mBCC cohort were analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 200 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
- LDE225 800mg mBCC: The efficacy and safety of LDE225 800mg mBCC cohort were analyzed separately in each group. Patients who met all the inclusion and none of the exclusion criteria were treated with 800 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Percentage of participants | 42.9 [27.7 to 59.0] | 37.6 [27.8 to 48.3] | 15.4 [1.9 to 45.4] | 17.4 [5.0 to 38.8]

2. Primary Outcome: Objective Response Rate (ORR) Based on Central Review According to mRECIST (for Locally Advanced Basal Cell Carcinoma (laBCC)) and RECIST 1.1 (Metastatic Basal Cell Carcinoma (mBCC)) Per Full Analysis Set (FAS)
Description: ORR is the percentage of patient's objective response (ORR) by 6 months after starting LDE225 treatment. A responder was defined as a subject with confirmed partial response (PR) or confirmed complete response (CR) 6 months after starting LDE225 treatment.Treatment with sonidegib was to be considered sufficiently efficacious if the observed ORR on any treatment arm at the end of the study was 30% or higher. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 6 months
Population: The full analysis set (FAS) comprised all patients who were assigned study treatment irrespective of receiving it (all randomized patients).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Percentage of participants | 47.0 [34.6 to 59.7] | 35.2 [26.9 to 44.1] | 15.4 [1.9 to 45.4] | 17.4 [5.0 to 38.8]

3. Secondary Outcome: Duration of Response (DoR) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: Duration of response is the time from the first observed confirmed response (CR or PR) to disease progression or death due to any reason.
  Duration of response was for participants with ORR. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  Progressive disease (PD): At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm2.
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 12.9 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 23.7 [10.8 to 29.6] | 24.0 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | NA [NA to NA] — N/A = Median DoR was non-estimable for patients with mBCC receiving treatment with sonidegib 800 mg as limited numbers of PD or death were observed.

4. Secondary Outcome: Duration of Response (DoR) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (FAS)
Description: Duration of response is the time from the first observed confirmed response (CR or PR) to disease progression or death due to any reason.
  Median DoR for patients with laBCC was non-estimable for both treatment arms. Duration of response was for participants with ORR. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Months | 26.1 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 23.3 [12.2 to 29.6] | 24.0 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | NA [NA to NA] — NA = Median DoR was non-estimable for patients with mBCC receiving treatment with sonidegib 800 mg as limited numbers of PD or death were observed.

5. Secondary Outcome: Complete Response Rate (CRR) Per Central Review (pEAS)
Description: Rate of complete response is the percentage of patients with best overall response of complete response (CR) after starting LDE225 treatment. The rate of CR was determined according to mRECIST for laBCC and RECIST 1.1 for mBCC. Patients with best overall response of 'Unknown" were treated as non responders. Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Percentage of participants | 4.8 [0.6 to 16.2] | 2.2 [0.3 to 7.6] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 14.8]

6. Secondary Outcome: Complete Response Rate (CRR) Per Central Review (FAS)
Description: Rate of complete response is the proportion of patients with best overall response of complete response (CR) after starting LDE225 treatment. The rate of CR will be determined according to mRECIST for laBCC and RECIST 1.1 for mBCC. Patients with best overall response of 'Unknown" will be treated as non responders
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Percentage of participants | 3.0 [0.4 to 10.5] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 14.8]

7. Secondary Outcome: Progression-free Survival (PFS) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: Progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 19.0 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 19.4 [13.8 to 30.5] | 13.1 [5.6 to 33.1] | 11.1 [7.3 to 16.6]

8. Secondary Outcome: Progression-free Survival (PFS) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (FAS)
Description: Progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
Time Frame: 42 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Months | 22.1 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 24.9 [19.2 to 33.4] | 13.1 [5.6 to 33.1] | 11.1 [7.3 to 16.6]

9. Secondary Outcome: Time to Tumor Response (TTR) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: Time to tumor response (TTR) is defined as the time from date of enrollment to the date of first documented tumor response (CR or PR). PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 4.0 [3.7 to 5.6] | 3.7 [2.0 to 5.5] | 9.2 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 1.0 [1.0 to 2.1]

10. Secondary Outcome: Time to Tumor Response (TTR) Per Central Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (FAS)
Description: as for outcome 9
Time Frame: 42 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 4.0 [3.7 to 5.6] | 3.7 [2.0 to 5.5] | 9.2 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed. | 1.0 [1.0 to 2.1]

11. Secondary Outcome: Objective Response Rate (ORR) Based on Site Investigator Review According to mRECIST (for Locally Advanced Basal Cell Carcinoma (laBCC)) and RECIST 1.1 (for Metastatic Basal Cell Carcinoma (mBCC)) Per Primary Efficacy Analysis Set (pEAS)
Description: ORR is the percentage of patient's objective response (ORR) by 42 months after starting LDE225 treatment. A responder was defined as a subject with confirmed partial response (PR) or confirmed complete response (CR) 42 months after starting LDE225 treatment. Treatment with sonidegib was considered sufficiently efficacious if the observed ORR on any treatment arm at the end of the study was 30% or higher. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Percentage of participants | 71.4 [55.4 to 84.3] | 61.3 [50.6 to 71.2] | 23.1 [5.0 to 53.8] | 34.8 [16.4 to 57.3]

12. Secondary Outcome: Objective Response Rate (ORR) Based on Site Investigator Review According to mRECIST (for Locally Advanced Basal Cell Carcinoma (laBCC)) and RECIST 1.1 (Metastatic Basal Cell Carcinoma (mBCC)) Per Full Analysis Set (FAS)
Description: ORR is the percentage of patient's objective response (ORR) by 6 months after starting LDE225 treatment. A responder was defined as a subject with confirmed partial response (PR) or confirmed complete response (CR) 42 months after starting LDE225 treatment.Treatment with sonidegib was to be considered sufficiently efficacious if the observed ORR on any treatment arm at the end of the study was 30% or higher. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Percentage of participants | 71.2 [58.7 to 81.7] | 58.6 [49.6 to 67.2] | 23.1 [5.0 to 53.8] | 34.8 [16.4 to 57.3]

13. Secondary Outcome: Duration of Response (DoR) Per Site Investigator Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: as for outcome 3
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 18.2 [12.9 to 23.0] | 26.0 [15.7 to 47.3] | 18.1 [17.7 to 18.4] | 10.2 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed.

14. Secondary Outcome: Duration of Response (DoR) Per Site Investigator Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (FAS)
Description: Duration of response is the time from the first observed confirmed response (CR or PR) to disease progression or death due to any reason. Duration of response was for participants with ORR. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: 42 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Months | 15.7 [12.0 to 20.2] | 26.0 [18.3 to 47.3] | 18.1 [17.7 to 18.4] | 10.2 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited numbers of PD or death were observed.

15. Secondary Outcome: Progression-free Survival (PFS) Per Site Investigator Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: as for outcome 7
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 20.1 [14.8 to 23.8] | 28.0 [19.4 to 49.8] | 13.1 [9.2 to 19.4] | 14.3 [11.1 to 17.0]

16. Secondary Outcome: Time to Tumor Response (TTR) Per Site Investigator Review Using mRECIST for laBCC and RECIST 1.1 for mBCC (pEAS)
Description: as for outcome 9
Time Frame: 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 42 | 93 | 13 | 23
Months | 1.9 [1.8 to 3.9] | 1.8 [1.1 to 2.0] | 1.0 [0.9 to 3.7] | 2.7 [1.0 to 5.6]

17. Secondary Outcome: Plasma Concentration of Sonidegib (LDE225)
Description: Blood PK samples were collected either by direct venipuncture or an indwelling cannula inserted in a forearm vein for the determination of trough (Cmin) plasma concentrations of sonidegib and its main circulating metabolite, LGE899, from all patients who enrolled in the study. Blood was collected in Weeks 1, 3, 5, 9 (pre-dose), and subsequently pre-dose every 4 weeks up to Week 21, and every 12 weeks thereafter up to week 69.
Time Frame: Weeks 1, 3, 5, 9, 13, 17, 21, 33, 45, 57, 69
Population: The PK analysis set (PAS) consisted of all patients with at least one evaluable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LDE225 200 mg qd: Patients who met all the inclusion and none of the exclusion criteria were treated with 200 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
- LDE225 800 mg qd: Patients who met all the inclusion and none of the exclusion criteria were treated with 800 mg LDE225 daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawal of consent.
Arm/Group | LDE225 200 mg qd | LDE225 800 mg qd
Number analyzed (Participants) | 73 | 139
ng/mL
  Week 1 (0 h (pre-dose)) | NA (NA) — N/A = Week1 pre-dose concentrations were below limit of quantitation | NA (NA) — N/A = Week1 pre-dose concentrations were below limit of quantitation
  Week 3 (0 h (pre-dose)): number analyzed (Participants) | 65 | 128
  Week 3 (0 h (pre-dose)) | 207.76 (78.29) | 586.76 (97.13)
  Week 5 (0 h (pre-dose)): number analyzed (Participants) | 70 | 120
  Week 5 (0 h (pre-dose)) | 372.26 (68.89) | 1012.63 (70.42)
  Week 9 (0 h (pre-dose)): number analyzed (Participants) | 68 | 101
  Week 9 (0 h (pre-dose)) | 559.29 (67.30) | 1353.06 (63.43)
  Week 13 (0 h (pre-dose)): number analyzed (Participants) | 63 | 85
  Week 13 (0 h (pre-dose)) | 714.01 (60.79) | 1443.84 (61.57)
  Week 17 (0 h (pre-dose)): number analyzed (Participants) | 66 | 81
  Week 17 (0 h (pre-dose)) | 688.93 (64.43) | 1574.21 (59.88)
  Week 17 (1 h (post-dose)): number analyzed (Participants) | 35 | 35
  Week 17 (1 h (post-dose)) | 841.78 (52.57) | 1803.74 (39.47)
  Week 17 (2 h (post-dose)): number analyzed (Participants) | 37 | 32
  Week 17 (2 h (post-dose)) | 939.56 (50.79) | 1922.38 (34.90)
  Week 17 (4 h (post-dose)): number analyzed (Participants) | 36 | 33
  Week 17 (4 h (post-dose)) | 842.31 (62.22) | 1750.70 (53.32)
  Week 17 (6 h (post-dose)): number analyzed (Participants) | 33 | 32
  Week 17 (6 h (post-dose)) | 759.88 (63.43) | 1673.95 (41.53)
  Week 21 (0 h (pre-dose)): number analyzed (Participants) | 58 | 67
  Week 21 (0 h (pre-dose)) | 707.49 (63.58) | 1547.41 (63.92)
  Week 33 (0 h (pre-dose)): number analyzed (Participants) | 49 | 49
  Week 33 (0 h (pre-dose)) | 702.67 (93.11) | 1477.60 (74.80)
  Week 45 (0 h (pre-dose)): number analyzed (Participants) | 33 | 35
  Week 45 (0 h (pre-dose)) | 697.92 (76.02) | 1368.87 (79.60)
  Week 57 (0 h (pre-dose)): number analyzed (Participants) | 22 | 26
  Week 57 (0 h (pre-dose)) | 559.17 (117.27) | 1257.42 (78.96)
  Wek 69 (0 h (pre-dose)): number analyzed (Participants) | 21 | 23
  Wek 69 (0 h (pre-dose)) | 530.91 (154.33) | 1355.91 (89.03)

18. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death due to any cause or the last date that a patient was known to be alive (censored observation) as of the data cut-off.
Time Frame: 42 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDE225 200mg laBCC | LDE225 800mg laBCC | LDE225 200mg mBCC | LDE225 800mg mBCC
Number analyzed (Participants) | 66 | 128 | 13 | 23
Months | NA [NA to NA] — N/A = Median OS was non-estimable for patients with laBCC receiving treatment with sonidegib 200 mg as limited number of deaths were observed. | NA [NA to NA] — N/A = Median OS was non-estimable for patients with laBCC receiving treatment with sonidegib 800 mg as limited number of deaths were observed. | 47.6 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited number of deaths were observed. | 33.8 [NA to NA] — N/A = Both lower and upper confidence intervals were not estimable as limited number of deaths were observed.

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 76.2 months.
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of approx. 7 years.
Arm/Group | LDE225 200 mg qd | LDE225 800 mg qd
All-Cause Mortality (participants affected / at risk) | 1/79 | 7/150
Serious Adverse Events (participants affected / at risk) | 16/79 | 58/150
Other Adverse Events (participants affected / at risk) | 76/79 | 145/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 200 mg qd (N=79) | LDE225 800 mg qd (N=150)
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4
Cardiac death (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pseudomonas infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 6
Lipase increased (Investigations) | 0 | 1
Myoglobin blood increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 5
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 200 mg qd (N=79) | LDE225 800 mg qd (N=150)
Anaemia (Blood and lymphatic system disorders) | 4 | 13
Vertigo (Ear and labyrinth disorders) | 0 | 11
Abdominal pain (Gastrointestinal disorders) | 8 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 12
Constipation (Gastrointestinal disorders) | 6 | 24
Diarrhoea (Gastrointestinal disorders) | 25 | 34
Dry mouth (Gastrointestinal disorders) | 4 | 8
Nausea (Gastrointestinal disorders) | 31 | 71
Vomiting (Gastrointestinal disorders) | 9 | 41
Asthenia (General disorders) | 10 | 9
Fatigue (General disorders) | 26 | 55
Pyrexia (General disorders) | 4 | 5
Influenza (Infections and infestations) | 4 | 8
Nasopharyngitis (Infections and infestations) | 8 | 17
Pneumonia (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 11
Urinary tract infection (Infections and infestations) | 7 | 7
Fall (Injury, poisoning and procedural complications) | 5 | 5
Blood creatine phosphokinase increased (Investigations) | 23 | 54
Lipase increased (Investigations) | 6 | 13
Weight decreased (Investigations) | 24 | 64
Decreased appetite (Metabolism and nutrition disorders) | 18 | 52
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 43 | 104
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 8
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Ageusia (Nervous system disorders) | 1 | 15
Dizziness (Nervous system disorders) | 7 | 15
Dysgeusia (Nervous system disorders) | 35 | 89
Headache (Nervous system disorders) | 12 | 20
Hypogeusia (Nervous system disorders) | 0 | 9
Paraesthesia (Nervous system disorders) | 4 | 6
Depression (Psychiatric disorders) | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 39 | 87
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 12
Hypertension (Vascular disorders) | 8 | 16

LIMITATIONS AND CAVEATS:
230 patients evaluated in the Full Analysis Set: 79 randomized to LDE225 (Sonidegib) 200mg group & 151 randomized to LDE225 800mg group. 1 patient randomized to the 800mg group did not receive study treatment & thus was not counted in the Safety Set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.